#### INFORMATION SHEET

Date: 2025-02-15

**Título del estudio:** Effectiveness of a multimodal intervention with simulation for learning home health nursing care of patients with multimorbidity and heart failure.

Principal Investigator: Antonio Jesús Marín Paz.

# INTRODUCTION

You are invited to participate in a study that has been approved by the Non-Animal Experimentation and Genetically Modified Organisms Ethics Committee (CEENB-OMGs) of the University of Cádiz, which is competent in non-clinical studies involving human subjects.

Please read this information sheet carefully. The researchers will clarify any questions you may have.

# **VOLUNTARY PARTICIPATION**

Your participation in this study is voluntary, and you may reverse your decision and withdraw your consent at any time.

# STUDY OVERVIEW

The objective of this project is to evaluate the efficacy of a multimodal intervention using high-fidelity simulations of home nursing visits in improving the care of multimorbid patients with heart failure.

To achieve this, we will ask you to complete a questionnaire requesting socio-demographic data, followed by questionnaires or scales related to learning and your experience with the simulation, as well as your level of satisfaction. In most cases, you will be asked to complete these on two occasions to assess the evolution of your nursing competencies and your experience in the simulations. Additionally, an alphanumeric code will be created for you to replace your full name on the questionnaires, enabling subsequent comparison of your data.

# BENEFITS AND RISKS OF PARTICIPATING IN THE STUDY

Participation in this project offers the benefit of more personalized learning regarding your performance in home nursing visits for the care of multimorbid patients with heart failure. There are no risks beyond those inherent in a typical educational simulation. To ensure that the educational research yields results consistent with its nature, it is essential that you maintain the confidentiality of the activities conducted during your individual simulation interventions and the teaching activities performed in the seminars.

#### FINANCIAL COMPENSATION

Your participation in this study will not incur any costs for you, nor will there be any financial compensation.

#### CONFIDENTIALITY

Your personal data collected during this study will be processed in accordance with the General Data Protection Regulation (GDPR) of the European Union and Organic Law 3/2018, of December 5, on Personal Data Protection and Guarantee of Digital Rights (LOPDGDD). Furthermore, you will be required to complete an audiovisual rights assignment document for the recording of simulation sessions and their subsequent processing for pedagogical purposes.

The purpose of processing personal data is to conduct research evaluating the efficacy of a multimodal intervention with high-fidelity simulations on home nursing visits to improve the care of multimorbid patients with heart failure. This research is coordinated by a nurse.

The data controller for personal data is Antonio Jesús Marín Paz. Contact details for the data controller for claims purposes are as follows: telephone: XXXXXXXX, email: XXXXXXX.

You may also contact us at the following postal address: Faculty of Nursing; Venus St., 11207 Algeciras, Cadiz, Spain.

Legal Basis: The processing of personal data is protected by the legal basis established in Articles 6.1.a) and 9.2.a) of the GDPR, which state that processing shall be lawful if the data subject or their legal representative has given explicit consent for the processing of their personal data for one or more specific purposes.

The data subject or their legal representative may grant consent for the use of their personal data for health research purposes, particularly biomedical research.

The purpose may encompass categories related to general areas linked to a medical or research specialty, all in accordance with Additional Provision Seventeenth 2.a) of the LOPDGDD.

Recipients or Categories of Recipients: Your personal data will be processed with the utmost confidentiality and will not be transferred to third parties unrelated to the research project. There are no other recipients or categories of recipients of your personal data. Under no circumstances will your personal data be subject to international data transfer. If the study results are published, your personal data will not be published, and your identity will remain anonymous.

# Exercise of Personal Data Protection Rights

You have the right to request from the data controller access to your personal data being processed. You also have the right to rectification of your personal data, to erasure of your personal data, to restriction of processing, to object to processing, to data portability, and not to be subject to decisions based solely on automated processing of your data. All of these rights are in accordance with and subject to the limitations set forth in the GDPR and the LOPDGDD for research purposes. These rights shall be exercised via the email address/postal address provided.

You may, at any time, exercise your right to withdraw consent for the processing of your personal and audiovisual data. This withdrawal will not affect the lawfulness of processing for educational research purposes based on consent given prior to its withdrawal. This right shall be exercised via the email address/postal address provided.

You have the right to lodge a complaint with the supervisory authority, which is the Andalusian Council for Transparency and Data Protection. This body exercises its jurisdiction over personal data processing managed by Andalusian regional institutions, the regional administration, local administrations, and other public and private entities dependent on any of these, as well as by universities within the Andalusian university system. For all other cases, you have the right to lodge a complaint with the Spanish Data Protection Agency.

# **FUNDING**

This study has no external funding sources.

#### WITHDRAWAL OF CONSENT

You may withdraw your consent at any time without needing to provide explanations, and without any academic consequences resulting from it. You should also be aware that you may be excluded from the study if the study investigators deem it appropriate.

You have the right to be informed of any changes to the study. In such a case, the investigator will need to request new consent from you, which you would be free to decline.

Before signing, please read this document carefully and ask any questions you deem appropriate after the research explanation. Should you have any doubts, please contact the principal investigator, Antonio Jesús Marín Paz.

#### Date: 2025-02-15

# WRITTEN INFORMED CONSENT

Study Title: Effectiveness of a multimodal intervention with simulation for learning home health nursing care of patients with multimorbidity and heart failure.

| I, (Participant's Full Name) |
|------------------------------|
|------------------------------|

- I have read and understood the information sheet provided to me.
- I have received sufficient information about the study.
- I understand that I must maintain the confidentiality of the study during its duration.
- I have had the opportunity to ask questions about the study.
- I understand that my participation is voluntary.
- I understand that I can withdraw from the study:
  - o At any time.
  - Without needing to provide explanations.
  - Without any academic repercussions in the course where this educational research will be conducted.

| Ιí | freely | give | my | conse | nt to | parti | cipate | in | this | stud | y. |
|---|---|---|---|---|---|---|---|---|---|---|---|

DATE:

PARTICIPANT'S SIGNATURE

# HOJA DE INFORMACIÓN

Fecha: 2025-02-15

**Título del estudio:** Efectividad de una intervención multimodal con simulación en paciente pluripatológicos con insuficiencia cardiaca en visita domiciliaria enfermera: ensayo aleatorio controlado

Investigador principal: Antonio Jesús Marín Paz

# INTRODUCCIÓN

Se le invita a participar en un estudio que ha sido aprobado por el Comité de Ética de Experimentación no animal y organismos modificados genéticamente (CEENB-OMGs) de la Universidad de Cádiz, competente en estudios no clínicos en los que seres humanos sean los sujetos de investigación.

Por favor, lea esta hoja informativa con atención. Los investigadores le aclararán las dudas que le puedan surgir.

# PARTICIPACIÓN VOLUNTARIA

Su participación en este estudio es voluntaria y usted puede anular su decisión y retirar el consentimiento en cualquier momento.

# DESCRIPCIÓN GENERAL DEL ESTUDIO

El objetivo del presente proyecto es evaluar la eficacia de una intervención multimodal con simulaciones de alta fidelidad sobre visitas domiciliarias enfermeras en la mejora de la atención de pacientes pluripatológicos con insuficiencia cardiaca.

Para ello, le solicitaremos que rellene un cuestionario donde se le solicitará la cumplimentación de datos sociodemográficos, y posteriormente cuestionarios o escalas relacionados con el aprendizaje y la experiencia a través de la simulación, así como el grado de satisfacción. En la mayoría de los casos, se le solicitará cumplimentarlos en dos ocasiones para comprobar la evolución de sus competencias enfermeras y de su experiencia en las simulaciones. Asimismo, se le creará un código alfanumérico en sustitución de su nombre y apellidos en los cuestionarios para poder realizar la comparación posteriormente.

# BENEFICIOS Y RIESGOS DERIVADOS DE SU PARTICIPACIÓN EN EL ESTUDIO

La participación en este proyecto supone el beneficio de un aprendizaje más personalizado en su grado de desempeño en las visitas domiciliarias enfermeras en el cuidado de pacientes pluripatológicos con insuficiencia cardíaca. No existen riesgos diferentes a los propios de una simulación docente habitual. Para garantizar que el desarrollo de la investigación docente

obtenga resultados acordes a la naturaleza del mismo, es esencial que usted mantenga la confidencialidad de la actividad realizada sobre sus intervenciones individuales de simulación y la actividad docente realizada en los seminarios.

# COMPENSACIÓN ECONÓMICA

Su participación en el estudio no supondrá ningún gasto para usted, ni existe compensación económica

# **CONFIDENCIALIDAD**

Sus datos personales recogidos en la realización de este estudio serán tratados según lo establecido en el Reglamento General de Protección de Datos de la Unión Europea (RGPD) y la Ley Orgánica 3/2018, de 5 de diciembre, de Protección de Datos de Carácter Personal y garantía de los derechos digitales (LOPDGDD). Asimismo, se le requerirá la cumplimentación de un documento de cesión de derechos audiovisuales para la grabación de las sesiones de simulación y su posterior tratamiento con fines pedagógicos.

La finalidad del tratamiento de los datos personales es la realización de una investigación para evaluar la eficacia de una intervención multimodal con simulaciones de alta fidelidad sobre visitas domiciliarias enfermeras en la mejora de la atención de pacientes pluripatológicos con insuficiencia cardiaca, cuya coordinación es ejercida por un enfermero.

Podrá dirigirse también a la siguiente dirección postal: Facultad de Enfermería; C/ Venus s/n, 11207 Algeciras, Cádiz, España.

Base legal: el tratamiento de datos personales se encuentra amparado en la base legal establecida en los arts. 6.1.a) y 9.2.a) del RGPD, que establece que el tratamiento será lícito si el interesado o su representante legal dio su consentimiento explícito para el tratamiento de sus datos personales para uno o varios fines específicos.

El interesado o su representante legal puede otorgar su consentimiento para el uso de sus datos personales con fines de investigación en salud, y, en particular, la biomédica.

La finalidad puede abarcar categorías relacionadas con áreas generales vinculadas a una especialidad médica o investigadora, todo ello de conformidad con la Disposición adicional decimoséptima 2.a) de la LOPDGDD.

Destinatarios o categorías de destinatarios. Sus datos personales serán tratados con la más absoluta confidencialidad por lo que no serán cedidos a terceras personas ajenas al proyecto de investigación. No existen destinatarios o categorías de destinatarios de sus datos personales. En ningún caso sus datos personales van a ser objeto de una transferencia internacional de datos personales. Si se publican los resultados del estudio, sus datos

personales no serán publicados y su identidad permanecerá anónima.

Ejercicio de los derechos de protección de datos personales

Tiene derecho a solicitar al responsable el acceso a sus datos personales sometidos a tratamiento. Asimismo, tiene derecho a la rectificación de sus datos personales, a la supresión de sus datos personales, a la limitación del tratamiento, a oponerse al tratamiento, a la portabilidad de los datos y, a no ser objeto de decisiones basadas únicamente en el tratamiento automatizado de sus datos, todo ello de conformidad y con las limitaciones previstas en el RGPD y en la LOPDGDD para la investigación. Estos derechos se ejercerán a través de la dirección de correo electrónico/dirección postal.

En cualquier momento puede ejercer el derecho a retirar el consentimiento para el tratamiento de sus datos personales y de derechos audiovisuales, sin que ello afecte a la licitud del tratamiento con fines de investigación docente basado en el consentimiento previo a su retirada. Este derecho se ejercerá a través de la dirección de correo electrónico/dirección postal.

Tiene el derecho a presentar una reclamación ante la autoridad de control, que es el Consejo de Transparencia y Protección de Datos Personales de Andalucía, que ejercer su competencia para los tratamientos de datos personales gestionados por las instituciones autonómicas de Andalucía, por la Administración autonómica, por las Administraciones locales, y por otras entidades de derecho público y privado dependientes de cualquiera de ellas, así como por las universidades del sistema universitario andaluz. Para el resto de los supuestos tiene el derecho a presentar una reclamación ante la Agencia Española de Protección de Datos.

# FINANCIACIÓN

Este estudio no dispone de ninguna fuente de financiación.

# RETIRADA DEL CONSENTIMIENTO

Usted puede retirar su consentimiento en cualquier momento sin tener que dar explicaciones, y sin que existan consecuencias académicas derivadas de ello. También debe saber que puede ser excluido del estudio si los investigadores del estudio lo consideran oportuno.

Usted tiene derecho a estar informado de cualquier cambio en el estudio. En ese caso, el investigador tendrá que pedirle un nuevo consentimiento que usted podría rechazar.

Antes de firmar, lea detenidamente el documento, haga todas las preguntas que considere oportunas tras la explicación de la investigación. En caso de duda debe dirigirse al investigador principal, Antonio Jesús Marín Paz.

Fecha: 2025-02-15

Título del estudio: Eficacia de una intervención multimodal con simulación en pacientes pluripatológicos con insuficiencia cardíaca en visita domiciliaria enfermera: ensayo controlado aleatorizado

CONSENTIMIENTO INFORMADO POR ESCRITO

| Yo (no | ombre y apellidos) |
|---|---|
| | He leído y comprendido la hoja de información que se me ha entregado. |
| | He recibido suficiente información sobre el estudio. |
| • | Comprendo que debo mantener la confidencialidad del estudio durante su periodo de realización. |

- He podido realizar preguntas sobre el estudio.
- Comprendo que mi participación es voluntaria.
- Comprendo que puedo retirarme del estudio:
  - o Cuando quiera.
  - o Sin tener que dar explicaciones.
  - Sin que ello repercuta, académicamente, en la asignatura donde se desarrollará la investigación docente.

| Presto libremente mi conformidad para participar en el estudio. |
|-----------------------------------------------------------------|
| FECHA: |

FIRMA DEL PARTICIPANTE